CLINICAL TRIAL: NCT05407103
Title: The Impact of Applying Various Forms of Acupressure on Women's Hand During Labor on Their Childbirth Comfort: A Randomized Controlled Trial
Brief Title: Acupressure and Comfort at Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serap Ozturk Altinayak (Other)
Responsible Party: Sponsor-Investigator, Serap Ozturk Altinayak, Assistant professor, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21.05.2020-15
Record Dates: First submitted 2022-05-29; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Pain, Labor
Keywords: Pain, Labor, Comfort
MeSH Terms: conditions — Labor Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cold Acupressure Group (Experimental): Personal information form (PIF ) , Labor Monitoring Form (LMF), Visual Analog Scale (VAS), and Childbirth Comfort Questionnaire (CCQ) as pre-test during the latent phase before going about the cold acupressure. Next, she applied the cold acupressure pouches on the respective cold group on their LI 4 point for ten minutes, during the active and transition phases. The application was then suspended for one hour, and then repeated three more times.
  Last, posttest took place. Cold group was given VAS and CCQ during transition phase of dilation between contractions. The researchers then filled out LMF after cold group to monitor how they were feeling.
  Interventions: Other: Cold Acupressure
- Warm Acupressure Group (Experimental): PIF, LMF, VAS, and CCQ as pre-test during the latent phase before going about the warm acupressure. Next, she applied the warm acupressure pouches on the respective warm groups on their LI 4 point for ten minutes, during the active and transition phases. The application was then suspended for one hour, and then repeated three more times.
  Last, posttest took place. Warm group was given VAS and CCQ during transition phase of dilation between contractions. The researchers then filled out LMF after warm group to monitor how they were feeling.
  Interventions: Other: Warm Acupressure
- Control Group (No Intervention): The researcher ran PIF, LMF, VAS, and CCQ as pre-test during the latent phase. No intervention was applied to the control group. Last, posttest took place. Control group was given VAS and CCQ during transition phase of dilation between contractions. The researchers then filled out LMF after warm group to monitor how they were feeling.

INTERVENTIONS:
Other: Cold Acupressure — For the cold acupressure application, the researchers prepared pouches that were 3 cm long, 2 cm wide, and 1 cm high (3x2x1cm), and filled with cherry seeds - to retain heat for a longer time, hence the preference. Next, they fixed rubber bands to the pouches so that they stayed in place on the participants' hands during acupressure, and retain consistent pressure throughout. Lastly, the cold acupressure pouches were kept in a freezer for 40 minutes.
  Arms: Cold Acupressure Group
Other: Warm Acupressure — For the warm acupressure application, the researchers prepared pouches that were 3 cm long, 2 cm wide, and 1 cm high (3x2x1cm), and filled with cherry seeds - to retain heat for a longer time, hence the preference. Next, they fixed rubber bands to the pouches so that they stayed in place on the participants' hands during acupressure, and retain consistent pressure throughout. Lastly, the warm acupressure pouches were heated in a microwave at 600 W for one minute.
  Arms: Warm Acupressure Group

SUMMARY:
Aims: Non-pharmacological methods employed for management labor pain also help pregnant women to cope with labor pain and increase their childbirth comfort. The aim of this study is to determine the effect of cold and hot acupressure applications, applied to the acupressure point LI4 of primiparous women during labor, on their childbirth comfort.

Methods: This study was designed a randomized controlled experimental study. The sample consisted of 129 healthy pregnant women including 44 pregnant women in the hot acupressure group, 44 pregnant women in the cold acupressure group, and 41 pregnant women in the control group. The "Personal Information Form", the "Labor Monitoring Form", the "Visual Analog Scale", and the "Childbirth Comfort Questionnaire" were all used to gather the data.

ELIGIBILITY:
Inclusion Criteria:

* Being a primipara
* Having intact membranes
* No skin diseases (such as urticaria...),
* No use of narcotic drugs
* Having a term pregnancy
* Having a single fetus at vertex position
* Planning to have vaginal delivery
* Having contractions and ongoing regular augmentation
* Having recent augmentation starting periods
* Being in the latent phase (0-3 cm dilatation)
* Having no history of high-risk pregnancy
* Not using analgesic drugs to reduce pain during delivery
* Having no systemic and neurologic diseases
* Having no contraction anomaly (hypotonic or hypertonic contractions)

Exclusion Criteria:

• Having any of the above criteria

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 129 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Comfort | through study completion, an average of 1month
  Childbirth Comfort Questionnaire (CCQ); Each item ranks between 1 and 5 points: 1=Strongly disagree, 2=Mostly disagree, 3=Partially agree, 4=Mostly agree, and 5=Completely agree. Thus, the lowest and highest scores are 9 and 45 points, respectively. The higher the score one earns, the more comfortable they are; the lower the score, the exact opposite

SECONDARY OUTCOMES:
Labor pain | through study completion, an average of 1month
  Visual Analog Scale (VAS); It is a 10-cm one-dimensional ruler; written on one end is "no pain"; on the other is "worst pain." For the purpose of this study, the researchers used VAS vertically in this study, in line with the recommendations of other studies, who suggest that individuals understand VAS better when applied vertically.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Research and Training Hospital of Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No